CLINICAL TRIAL: NCT06023654
Title: Preliminary Validation of a Novel Screening Tool and Diagnostic Criteria to Identify Circadian Rest-Activity Rhythm Disorders in Patients With Advanced Cancer
Brief Title: Identifying Circadian Rest-Activity Rhythm Disorders in Patients With Advanced Cancer
Status: Completed | Type: Observational
Sponsor: University of Dublin, Trinity College (Other)
Collaborators: Our Lady's Hospice and Care Services (Other)
Responsible Party: Principal Investigator, Prof Andrew Davies, Professor of Palliative Medicine, University of Dublin, Trinity College
Other Study IDs: 1926A
Record Dates: First submitted 2022-09-09; First posted 2023-09-05 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Cancer; Circadian Rhythm Disorders; Sleep Disturbance; Activity, Motor; Accelerometry
MeSH Terms: conditions — Neoplasms; Chronobiology Disorders; Parasomnias; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Circadian rest-Activity Rhythm disorders (CARDs) are common in patients with cancer, particularly in advanced disease. CARDs are associated with increased symptoms, poorer quality of life, poorer response to anticancer treatments and shorter survival.

The goal of this observational study is to see how common CARDs are in patients with advanced cancer and to characterise their rest and activity patterns in more detail.

A recent study has outlined a standard way to assess and diagnose a CARD.

This study aims to assess patients with advanced cancer for a CARD using a novel screening tool against this newly formed diagnostic criteria. Potentially modifiable risk factors will be considered along with associations between CARDs and symptoms, sleep preferences, sleep quality, daytime sleepiness, quality of life measures and predictors of survival.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years of age or older)
* Locally advanced or metastatic cancer
* Outpatient
* Ambulatory
* Prognosis of 3 months or more

Exclusion Criteria:

* Inpatient
* Shiftworker
* Recent long-haul travel
* Cognitive impairment impacting on ability to complete questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced or metastatic cancer
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-22 (Actual)

PRIMARY OUTCOMES:
To measure preliminary concurrent validity of a novel screening tool to identify Circadian rest-Activity Rhythm Disorders in patients with advanced cancer against diagnostic criteria | Time 1 (baseline), Time 2 (after 72 consecutive hours of accelerometry monitoring)
  Assessing the sensitivity and specificity of the screening tool

SECONDARY OUTCOMES:
To measure test-retest reliability of a novel screening tool to identify Circadian rest-Activity Rhythm Disorders in patients with advanced cancer | Time 1 (baseline), Time 2 (after 72 consecutive hours of accelerometry monitoring)
  Assessing the correlation between scores from the screening tool at two time points
To measure acceptability and ease of use of a novel screening tool to identify Circadian rest-Activity Rhythm Disorders in patients with advanced cancer | Time 2 (after 72 consecutive hours of accelerometry monitoring)
  Patient ease of use, understandability, acceptability and time to complete.
To measure acceptability and ease of use of a novel sleep and activity diary in patients with advanced cancer | Time 2 (after 72 consecutive hours of accelerometry monitoring)
  Patient ease of use, understandability, and acceptability
To identify the incidence of Circadian rest-activity Rhythm Disorders in patients with advanced cancer | Time 2 (after 72 consecutive hours of accelerometry monitoring)
  Incidence of Circadian rest-Activity Rhythm Disorders as identified by diagnostic criteria
To assess rest and physical activity patterns in patients with advanced cancer | Time 2 (after 72 consecutive hours of accelerometry monitoring)
  Combined assessment using wrist and thigh accelerometry alongside a sleep and activity diary
To assess the relationship between demographic details and the risk of developing a Circadian rest-Activity Rhythms in patients with cancer | Time 2 (after 72 consecutive hours of accelerometry monitoring)
  Baseline demographic details collected using a questionnaire
To assess the relationship between past medical history and the risk of developing a Circadian rest-Activity Rhythms in patients with cancer | Time 2 (after 72 consecutive hours of accelerometry monitoring)
  Past medical history collected using a questionnaire
To assess the relationship between current medication use and the risk of developing a Circadian rest-Activity Rhythms in patients with cancer | Time 2 (after 72 consecutive hours of accelerometry monitoring)
  Current medication use collected using a questionnaire
To assess the relationship between chronotype and the risk of develop a Circadian rest-Activity Rhythms in patients with cancer | Time 2 (after 72 consecutive hours of accelerometry monitoring)
  Chronotype assessed using the Morningness-Eveningness Questionnaire (MEQ)
To assess the relationship between occupation and the risk of developing a Circadian rest-Activity Rhythms in patients with cancer | Time 2 (after 72 consecutive hours of accelerometry monitoring)
  Occupation provided by participant using a questionnaire
To assess the relationship between cigarette use and the risk of developing a Circadian rest-Activity Rhythms in patients with cancer | During 72 hours period of monitoring
  Number and timing of last cigarette smoked each day assessed using a patient diary
To assess the relationship between alcohol consumption and the risk of developing a Circadian rest-Activity Rhythms in patients with cancer | During 72 hours period of monitoring
  Number and timing of alcoholic beverages consumed each day assessed using a patient diary
To assess the relationship between caffeine consumption and the risk of developing a Circadian rest-Activity Rhythms in patients with cancer | During 72 hours period of monitoring
  Number and timing of last of caffeinated drink consumed each day assessed using a patient diary
To assess associations between Circadian rest-activity Rhythm Disorders in patients with advanced cancer with symptoms | Time 2 (after 72 consecutive hours of accelerometry monitoring)
  Symptoms measured using the Memorial Symptom Assessment Scale - Short Form (MSAS-SF)
To assess associations between Circadian rest-activity Rhythm Disorders in patients with advanced cancer and prognosis | Time 2 (after 72 consecutive hours of accelerometry monitoring)
  Prognosis measured using the Prognosis in Palliative Care tool (PiPS-B)
To assess associations between Circadian rest-activity Rhythm Disorders in patients with advanced cancer with quality of life | Time 2 (after 72 consecutive hours of accelerometry monitoring)
  Quality of Life measured using the EORTC Quality of Life Questionnaire (EORTC-QLQ-C30)
To assess associations between Circadian rest-activity Rhythm Disorders in patients with advanced cancer with sleep quality | Time 2 (after 72 consecutive hours of accelerometry monitoring)
  Sleep quality measured using the brief Pittsburgh Sleep Quality Instrument (bPSQI)
To assess associations between Circadian rest-activity Rhythm Disorders in patients with advanced cancer with daytime sleepiness | Time 2 (after 72 consecutive hours of accelerometry monitoring)
  Daytime sleepiness assess using the Epworth Sleepiness Scale

CONTACTS AND LOCATIONS:
Locations (2):
- Ireland (2):
  - Our Lady's Hospice & Care Services, Dublin
  - St James's Hospital, Dublin